CLINICAL TRIAL: NCT06483529
Title: Respiratory Mechanics Measurement of Ventilated Patients Through Low-frequency Oscillometry Technique, an Explorative Study
Brief Title: Respiratory Mechanics Measurement of Ventilated Patients Through Low-frequency Oscillometry Technique
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: EC-2023-188-MDR
Record Dates: First submitted 2023-09-27; First posted 2024-07-03 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Ventilator Lung
Keywords: oscillometry; intensive care unit; intubated patients; compliance; resistance; impedance
MeSH Terms: conditions — Patient Compliance

STUDY DESIGN:
Intervention Model Description: prospective equivalence study with a two-arm crossover design - explorative pilot study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- ROELEC PROTOCOL (Experimental): ROELEC measurements consist of the application of a sine or multisine excitation pressure signal superimposed on the ventilation signal. The novelties are in the smart design of the excitation signal, not the way it is applied to the patient.
  Interventions: Diagnostic Test: compliance measurement
- dynamic P/V curves (Active Comparator): dynamic ventilatory pressure volume curves generated during the standard ventilation settings
  Interventions: Diagnostic Test: compliance measurement
- low flow P/V curves (Other): static ventilatory pressure volume curves will be generated during the procedure to assure that the patients ventilation is between the lower inflection point and the higher inflection point. this P/V curves will also be analysed but will not be included in the primary endpoint analysis
  Interventions: Diagnostic Test: compliance measurement
- SOTA (Other): Standard of care oscillometry protocol will also generate low flow P/V curves but will not be included in the primary endpoint analysis
  Interventions: Diagnostic Test: compliance measurement

INTERVENTIONS:
Diagnostic Test: compliance measurement — compliance can be measured by analyzing pressure volume curves generated through different methods

SUMMARY:
Respiratory failure has historically been one of the most important causes for admittance of patients to the critical care unit. This problem was the most important reason during the COVID-19 pandemic. Following the evolution of the physiology of the lung has therefore been the number one concern during these challenging times in the intensive care unit (ICU). Respiratory oscillometry (RO) identifies the lung impedance by applying small pressure oscillations onto the breathing or ventilation. Information about the respiratory mechanics can be extracted out of this impedance, including the resistance (R) and compliance (C) of the lung. The VUB developed a robust, patient safe RO measurement protocol that delivers high quality measurements with the least possible interference with the patient's breathing/ventilation. The technique challenges current state-of-the-art techniques also aiming at identifying R and C of the respiratory system (not exclusively RO). The RO measurement protocol is in line with the technical standards of the ERS (European Respiratory Society) and has been successfully and safely tested on emulators and some parts on test subjects. The clinical investigation aims at a powered equivalence investigation between the RO measurement protocol and a standard of care dynamic compliance estimate on invasive ventilated patients. As secondary objectives, the feasibility of the RO techniques will be investigated during pressure support ventilation and the RO estimates will also be compared with other accepted respiratory mechanics estimation tools. To enable the investigation, a RO algorithm is developed, and a RO measurement extension is implemented in the DemcAir® ventilation system of Demcon. This was a fully tested ventilator that received a CE mark under the previous MDD regulation. However, Demcon, which produces ventilator parts for other commercial partners, removed the label to avoid competition with their partners. The ventilator will only execute the protocol on demand and save the data on an USB stick available in the ventilator. At any time, the RO measurement procedure can be stopped, and the ventilator will return to its initial ventilation. The USB stick is used to transport the data to a separate (VUB) laptop where the data processing is done.

ELIGIBILITY:
Inclusion Criteria:

* intubation
* Controlled ventilation with an intention to continue controlled ventilation for the following 4 hours.
* Richmond agitation sedation scale of -4 or less
* Hemodynamically stable patient with either

  * unchanged vasopressor dose administration for at least 60 minutes before the start of the measurements
  * no vasopressor need and no vasopressor initiated within 60 minutes of measurements
* No planned intervention in the coming 2 hours
* Survival for at least 48 hours
* Protective ventilation (inspired oxygen concentration≤60%, plateau pressure ≤30 cmH2O , driving pressure≤ 15cmH2O)
* PEEP (Positive End Expiratory Pressure) ≤10

Exclusion Criteria:

* assist ventilation
* Ventilator asynchronies
* Intermittent spontaneous breathing
* nitric oxide therapy
* presence of an extra corporeal membrane oxygenation device
* Ventilation is not possible within the lower and upper inflection point of the low flow pressure volume curve.
* Unstable right heart failure
* Unstable lung embolism
* Standard of care without Sedline® or invasive arterial catheter
* Do not reanimate code of 2, 3 or 4
* Subjects who are healthy, minors, pregnant women, patients in emergency situation
* Outside the age range 18 to 84 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2023-09-18 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
compliance | Twice a day with at least 4hour interval, during 1 hour, compliance will be measured in every interventional action: ROELEC protocol, SOTA, dynamic P/V curve and low flow P/V curve
  compliance of the lung expressed in "ml/cmH20 "

SECONDARY OUTCOMES:
resistance | Twice a day with at least 4hour interval, during 1 hour, resistance will be measured in every interventional action: ROELEC protocol, SOTA, dynamic P/V curve and low flow P/V curve
  resistance of the lung expressed in cmH20/L/sec
impedance | Twice a day with at least 4hour interval, during 1 hour, impedance will be measured in every interventional action: ROELEC protocol, SOTA, dynamic P/V curve and low flow P/V curve
  lung impedance expressed in Ohm

CONTACTS AND LOCATIONS:
Overall Officials: joop jonckheer, MD, PhD, Principal Investigator — Universitair Ziekenhuis Brussel
Locations (1):
- Universitair Ziekenhuis Brussel, Jette, Brussel Hoofstedelijk Gewest, Belgium

IPD SHARING:
Plan to Share IPD: Yes
The Clinical Trial Summary Excel file and the .mat files can be shared safely on a request basis, given the anonymization scheme. This will allow other researchers to run their processing on the dataset and reach their own conclusions.
  The GDPR additional Excel file, or Mapping Table, and the eCRF will never be shared with anyone outside the principal investigator/authorized study member. With it, anyone can identify the patients who took part in the clinical trial.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: after the most important manuscript(s) will be published, data will be shared. however upon request for review of the manuscript data can be shared.
Access Criteria: after the most important manuscript(s) will be published, data will be shared. however upon request for review of the manuscript data can be shared.